CLINICAL TRIAL: NCT03695237
Title: A Phase 3, Multicenter, Open-Label, Two-Part Study to Evaluate the Safety, Efficacy, Pharmacokinetics, and Pharmacodynamics of Leuprolide Acetate 45 mg 6-Month Depot Formulation in Children With Central Precocious Puberty (CPP)
Brief Title: A Study to Evaluate Leuprolide Acetate 45 mg 6-Month Formulation in Children With Central Precocious Puberty (CPP)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M16-904
Record Dates: First submitted 2018-10-02; First posted 2018-10-04 (Actual); Results first posted 2023-05-16 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Central Precocious Puberty (CPP)
Keywords: Central Precocious Puberty (CPP); Leuprolide Acetate (LA)
MeSH Terms: conditions — Puberty, Precocious | interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Leuprolide Acetate (LA) (Experimental): Participants received leuprolide acetate (LA) 45 mg every 6 months administered as an intramuscular injection for up to 144 weeks.
  Interventions: Drug: Leuprolide Acetate (LA)

INTERVENTIONS:
Drug: Leuprolide Acetate (LA) — Administered intramuscularly as an injection
  Other Names: Lupron Depot

SUMMARY:
The primary objective of the study is to assess the safety and efficacy of a leuprolide acetate (LA) 45 mg 6-month depot formulation for the treatment of CPP in children who are either naïve to treatment with a gonadotropin-releasing hormone agonist (GnRHa) or who have been previously treated with a GnRHa.

ELIGIBILITY:
Inclusion Criteria:

* Children with CPP who are naïve to treatment with a gonadotropin-releasing hormone agonist (GnRHa) (females 2 - 8 years of age, or males 2 - 9 years of age) or who have been on standard GnRHa therapy for at least 6 months (females 2 - 10 years of age, or males 2 - 11 years of age).
* No history of clinically significant medical conditions or any other reason that the investigator determines would make the participant an unsuitable candidate to receive study drug.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2018-10-24 (Actual); Primary Completion 2021-05-06 (Actual); Study Completion 2023-11-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (18):
- United States (17):
  - Pediatric Endocrinology Associates /ID# 200629, Long Beach, California
  - Rady Children's Hospital San Diego /ID# 202491, San Diego, California
  - Children's Hospital Colorado /ID# 201645, Aurora, Colorado
  - Pediatric Endocrine Associates /ID# 201089, Greenwood Village, Colorado
  - Nemours Children's Health System /ID# 201331, Jacksonville, Florida
  - Arnold Palmer Hospital /ID# 201624, Orlando, Florida
  - Van Meter Pediatric Endocrinology /ID# 201688, Atlanta, Georgia
  - Rocky Mountain Diabetes and Osteoporosis Center /ID# 209878, Idaho Falls, Idaho
  - Indiana University /ID# 200526, Indianapolis, Indiana
  - Pediatric Endocrine Associates /ID# 202396, Boston, Massachusetts
  - University of Minnesota /ID# 200508, Minneapolis, Minnesota
  - Children's Mercy Hospital/ID# 200221, Kansas City, Missouri
  - University of Oklahoma /ID# 200659, Tulsa, Oklahoma
  - Penn State Hershey Medical Ctr /ID# 200287, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia - Main /ID# 203846, Philadelphia, Pennsylvania
  - Cook Children's Med. Center /ID# 212937, Fort Worth, Texas
  - Multicare Institute for Research and Innovation /ID# 202188, Tacoma, Washington
- Pediatric Endocrine Research Associates /ID# 200131, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 16 sites in the United States including Puerto Rico.
  The study enrolled pediatric participants with central precocious puberty (CPP) who were either naïve to treatment with a gonadotropin-releasing hormone receptor agonist (GnRHa) or who had been previously treated with a GnRHa.
Pre-assignment Details: The study was conducted in 2 parts. In Part 1, leuprolide acetate (LA) 45 mg 6-month depot formulation was evaluated from Baseline to Week 48. Following completion of Part 1 assessments, participants continued in Part 2 (extension period) to evaluate long-term treatment of LA 45 mg 6-month depot formulation (up to 24 months).
Groups:
- Leuprolide Acetate - Previously Treated: Participants who had been previously treated with a GnRHa for at least 6 months prior to enrollment received leuprolide acetate (LA) 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1 and for up to an additional 96 weeks in Part 2.
- Leuprolide Acetate - Treament Naïve: Participants without previous GnRHa treatment prior to enrollment (treatment naïve) received leuprolide acetate 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1 and for up to an additional 96 weeks in Part 2.
Period: Overall Study
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve
Started | 18 | 27
Completed | 8 | 20
Not Completed | 10 | 7
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Lost to Follow-up | 1 | 2
Not completed — Other, Not Specified | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Leuprolide Acetate - Previously Treated: Participants who had been previously treated with a GnRHa for at least 6 months prior to enrollment received leuprolide acetate (LA) 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1.
- Leuprolide Acetate - Treament Naïve: Participants without previous GnRHa treatment prior to enrollment (treatment naïve) received leuprolide acetate 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1.
- Total: Total of all reporting groups
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Total
Number analyzed (Participants) | 18 | 27 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.1 (1.73) | 7.7 (0.83) | 7.8 (1.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 24 | 41
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 9 | 11
  Not Hispanic or Latino | 16 | 18 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 12 | 18 | 30
  More than one race | 0 | 6 | 6
  Unknown or Not Reported | 0 | 0 | 0
Age at onset of CPP [Mean (Standard Deviation); unit: years] — Population: Reported by sex and overall
  years
    Females: number analyzed (Participants) | 17 | 24 | 41
    Females | 5.9 (2.37) | 6.7 (0.99) | 6.4 (1.74)
    Males: number analyzed (Participants) | 1 | 3 | 4
    Males | 2.1 | 6.9 (2.58) | 5.7 (3.19)
    Overall | 5.7 (2.46) | 6.8 (1.18) | 6.3 (1.86)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Suppression of Peak Gonadotropin-releasing Hormone Agonist (GnRHa)-Stimulated Luteinizing Hormone (LH) to Less Than 4 mlU/mL at Week 24
Description: Suppression of GnRHa-stimulated luteinizing hormone (LH) was measured using a peak GnRHa stimulation test, performed using subcutaneous injection with an aqueous formulation of leuprolide acetate at 20 µg/kg.
  Peak stimulated LH was calculated by taking the maximum LH concentrations measured from blood samples taken at 30 or 60 min following the GnRHa stimulation test.
  Suppression of GnRHa-stimulated luteinizing hormone is defined as peak stimulated LH less than 4 mIU/mL.
Time Frame: Week 24 (prior to the Week 24 dose); samples for LH measurement were taken 30 and 60 minutes after the stimulation test injection.
Population: The Full Analysis Set (FAS) consists of all participants who received at least 1 dose of study drug. Participants with missing GnRHa-stimulated LH results at Week 24 were counted as not achieving suppression.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Leuprolide Acetate - Previously Treated: Participants who had been previously treated with a GnRHa for at least 6 months prior to enrollment received leuprolide acetate 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1.
- Leuprolide Acetate - Overall: Participants received leuprolide acetate 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1.
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 18 | 27 | 45
percentage of participants | 94.4 [72.7 to 99.9] | 81.5 [61.9 to 93.7] | 86.7 [73.2 to 95.0]

2. Secondary Outcome: Part 1: Percentage of Participants With Suppression of Peak GnRHa-stimulated LH to Less Than 4 mlU/mL at Weeks 12, 20, 44, and 48
Description: as for outcome 1
Time Frame: Weeks 12, 20, 44, and 48 (prior to Week 48 dose); samples for LH measurement were taken 30 and 60 minutes after the stimulation test injection.
Population: The Full Analysis Set (FAS) consists of all participants who received at least 1 dose of study drug. Participants with missing GnRHa-stimulated LH results at a specific visit were counted as not achieving suppression for that visit.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 18 | 27 | 45
percentage of participants
  Week 12 | 83.3 [58.6 to 96.4] | 88.9 [70.8 to 97.7] | 86.7 [73.2 to 95.0]
  Week 20 | 94.4 [72.7 to 99.9] | 85.2 [66.3 to 95.8] | 88.9 [76.0 to 96.3]
  Week 44 | 88.9 [65.3 to 98.6] | 88.9 [70.8 to 97.7] | 88.9 [76.0 to 96.3]
  Week 48 | 83.3 [58.6 to 96.4] | 92.6 [75.7 to 99.1] | 88.9 [76.0 to 96.3]

3. Secondary Outcome: Part 1: Percentage of Female Participants With Suppression of Basal Estradiol to < 20 pg/mL at Weeks 12, 20, 24, 44, and 48
Description: Estradiol concentrations were measured from blood samples taken at each study visit prior to stimulation testing (and prior to study drug administration at Weeks 24 and 48).
Time Frame: Weeks 12, 20, 24, 44, and 48
Population: Full analysis set; female participants with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 17 | 24 | 41
percentage of participants
  Week 12: number analyzed (Participants) | 16 | 22 | 38
  Week 12 | 100.0 [79.4 to 100.0] | 95.5 [77.2 to 99.9] | 97.4 [86.2 to 99.9]
  Week 20: number analyzed (Participants) | 16 | 23 | 39
  Week 20 | 100.0 [79.4 to 100.0] | 95.7 [78.1 to 99.9] | 97.4 [86.5 to 99.9]
  Week 24: number analyzed (Participants) | 17 | 21 | 38
  Week 24 | 100.0 [80.5 to 100.0] | 95.2 [76.2 to 99.9] | 97.4 [86.2 to 99.9]
  Week 44: number analyzed (Participants) | 17 | 23 | 40
  Week 44 | 100.0 [80.5 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [91.2 to 100.0]
  Week 48: number analyzed (Participants) | 16 | 24 | 40
  Week 48 | 100.0 [79.4 to 100.0] | 100.0 [85.8 to 100.0] | 100.0 [91.2 to 100.0]

4. Secondary Outcome: Part 1: Percentage of Male Participants With Suppression of Basal Testosterone to < 30 ng/dL at Weeks 12, 20, 24, 44, and 48
Description: Testosterone concentrations were measured from blood samples taken at each study visit prior to stimulation testing (and prior to study drug administration for Weeks 24 and 48).
Time Frame: Weeks 12, 20, 24, 44, and 48
Population: Full analysis set; male participants with available data at each time point
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 1 | 3 | 4
percentage of participants
  Week 12: number analyzed (Participants) | 1 | 2 | 3
  Week 12 | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0]
  Week 20: number analyzed (Participants) | 1 | 2 | 3
  Week 20 | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0] | 100.0 [29.2 to 100.0]
  Week 24 | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [39.8 to 100.0]
  Week 44 | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [39.8 to 100.0]
  Week 48 | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [39.8 to 100.0]

5. Secondary Outcome: Parts 1 and 2: Percentage of Participants With Suppression of the Physical Signs of Puberty
Description: Breast development in females and testicular volume or genital development in males was assessed using modified Tanner staging, on a scale from Stage 1 (prepubertal) to Stage 5 (adult characteristics).
  Females: Suppression is defined as regression or no progression of breast development according to modified Tanner staging.
  Males: Suppression is defined as regression or no progression in testicular volume and genital staging according to modified Tanner staging.
Time Frame: Part 1: Weeks 24 and 48; Part 2: Weeks 72, 96, 120, and 144
Population: Full analysis set; results for males and females (with an assessment at each time point) are reported separately.
Measure: Number; unit: percentage of participants
Groups:
- Leuprolide Acetate - Previously Treated: Participants who had been previously treated with a GnRHa for at least 6 months prior to enrollment received leuprolide acetate 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1 and for up to an additional 96 weeks in Part 2.
- Leuprolide Acetate - Overall: Participants received leuprolide acetate 45 mg every 6 months administered as an intramuscular injection for up to 48 weeks in Part 1 and for up to an additional 96 weeks in Part 2.
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 18 | 27 | 45
percentage of participants
  Females: Week 24: number analyzed (Participants) | 17 | 24 | 41
  Females: Week 24 | 94.1 | 91.7 | 92.7
  Females: Week 48: number analyzed (Participants) | 17 | 24 | 41
  Females: Week 48 | 88.2 | 91.7 | 90.2
  Females: Week 72: number analyzed (Participants) | 16 | 23 | 39
  Females: Week 72 | 93.8 | 95.7 | 94.9
  Females: Week 96: number analyzed (Participants) | 14 | 21 | 35
  Females: Week 96 | 100 | 90.5 | 94.3
  Females: Week 120: number analyzed (Participants) | 12 | 19 | 31
  Females: Week 120 | 91.7 | 89.5 | 90.3
  Females: Week 144: number analyzed (Participants) | 6 | 16 | 22
  Females: Week 144 | 83.3 | 87.5 | 86.4
  Males: Week 24: number analyzed (Participants) | 1 | 3 | 4
  Males: Week 24 | 0 | 66.7 | 50.0
  Males: Week 48: number analyzed (Participants) | 1 | 3 | 4
  Males: Week 48 | 100 | 66.7 | 75.0
  Males: Week 72: number analyzed (Participants) | 1 | 3 | 4
  Males: Week 72 | 0 | 66.7 | 50.0
  Males: Week 96: number analyzed (Participants) | 1 | 3 | 4
  Males: Week 96 | 100 | 66.7 | 75.0
  Males: Week 120: number analyzed (Participants) | 1 | 3 | 4
  Males: Week 120 | 0 | 66.7 | 50.0
  Males: Week 144: number analyzed (Participants) | 1 | 1 | 2
  Males: Week 144 | 0 | 100 | 50.0

6. Secondary Outcome: Parts 1 and 2: Change From Baseline in Incremental Growth Rate
Description: Growth rate (height in centimeter/year) was calculated both prior to treatment in the study and during the study. For Baseline calculation a historical measurement of height at least 6 months prior to Screening and the Screening value was used.
Time Frame: Part 1: Baseline and Weeks 4, 12, 20, 24, 44, and 48; Part 2: Weeks 72, 96, 120, and 144
Population: Full analysis set; participants with available data at Baseline (43 participants) and each time point.
Measure: Mean (Standard Deviation); unit: cm/year
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 17 | 26 | 43
cm/year
  Week 4 | -0.6 (9.99) | -0.9 (10.52) | -0.8 (10.19)
  Week 12: number analyzed (Participants) | 16 | 25 | 41
  Week 12 | -0.6 (4.09) | -2.9 (5.42) | -2.0 (5.02)
  Week 20: number analyzed (Participants) | 16 | 24 | 40
  Week 20 | -0.5 (2.61) | -3.8 (4.69) | -2.5 (4.28)
  Week 24 | -0.5 (2.81) | -3.7 (4.28) | -2.4 (4.03)
  Week 44: number analyzed (Participants) | 17 | 25 | 42
  Week 44 | -0.4 (2.48) | -4.1 (3.77) | -2.6 (3.76)
  Week 48: number analyzed (Participants) | 16 | 26 | 42
  Week 48 | -0.3 (2.67) | -3.5 (4.71) | -2.3 (4.32)
  Week 72: number analyzed (Participants) | 16 | 25 | 41
  Week 72 | -0.5 (2.09) | -4.3 (3.53) | -2.8 (3.55)
  Week 96: number analyzed (Participants) | 15 | 23 | 38
  Week 96 | -0.6 (2.29) | -4.9 (3.43) | -3.2 (3.68)
  Week 120: number analyzed (Participants) | 13 | 21 | 34
  Week 120 | -1.2 (1.96) | -5.6 (3.27) | -3.9 (3.54)
  Week 144: number analyzed (Participants) | 7 | 16 | 23
  Week 144 | -1.0 (1.63) | -5.3 (2.76) | -4.0 (3.19)

7. Secondary Outcome: Parts 1 and 2: Ratio of Change From Baseline in Bone Age to Change From Baseline in Chronological Age
Description: Bone age was assessed from radiographs of the hand and wrist by a central imaging vendor using the BoneXpert automated system.
  A ratio less than 1 indicates less advancement of bone age compared to chronological age.
Time Frame: Part 1: Baseline and Weeks 24 and 48; Part 2: Weeks 72, 96, 120, and 144
Population: Full analysis set; based on non missing observations.
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 18 | 27 | 45
ratio
  Week 24 | 0.5 (0.80) | 0.7 (0.56) | 0.6 (0.66)
  Week 48 | 0.2 (1.36) | 0.6 (0.41) | 0.5 (0.93)
  Week 72: number analyzed (Participants) | 17 | 26 | 43
  Week 72 | 0.6 (0.31) | 0.6 (0.38) | 0.6 (0.35)
  Week 96: number analyzed (Participants) | 15 | 24 | 39
  Week 96 | 0.6 (0.32) | 0.7 (0.28) | 0.6 (0.29)
  Week 120: number analyzed (Participants) | 13 | 22 | 35
  Week 120 | 0.5 (0.28) | 0.6 (0.34) | 0.6 (0.32)
  Week 144: number analyzed (Participants) | 7 | 17 | 24
  Week 144 | 0.6 (0.26) | 0.6 (0.24) | 0.6 (0.24)

8. Secondary Outcome: Part 2: Percentage of Participants With Maintenance of Suppression of GnRHa-stimulated LH (< 4 mlU/mL)
Description: as for outcome 1
Time Frame: Weeks 72, 96, 120, and 144
Population: Full analysis set; observed cases.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 17 | 26 | 43
percentage of participants
  Week 72 | 88.2 [63.6 to 98.5] | 96.2 [80.4 to 99.9] | 93.0 [80.9 to 98.5]
  Week 96: number analyzed (Participants) | 15 | 23 | 38
  Week 96 | 93.3 [68.1 to 99.8] | 95.7 [78.1 to 99.9] | 94.7 [82.3 to 99.4]
  Week 120: number analyzed (Participants) | 13 | 22 | 35
  Week 120 | 100.0 [75.3 to 100.0] | 100.0 [84.6 to 100.0] | 100.0 [90.0 to 100.0]
  Week 144: number analyzed (Participants) | 7 | 16 | 23
  Week 144 | 100.0 [59.0 to 100.0] | 100.0 [79.4 to 100.0] | 100.0 [85.2 to 100.0]

9. Secondary Outcome: Part 2: Percentage of Female Participants With Maintenance of Suppression of Basal Estradiol to < 20 pg/mL
Description: Estradiol concentrations were measured from blood samples taken at each study visit prior to stimulation testing.
Time Frame: Weeks 72, 96, 120, and 144
Population: Full analysis set; participants with non-missing observations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 16 | 23 | 39
percentage of participants
  Week 72 | 100.0 [79.4 to 100.0] | 100.0 [85.2 to 100.0] | 100.0 [91.0 to 100.0]
  Week 96: number analyzed (Participants) | 14 | 20 | 34
  Week 96 | 100.0 [76.8 to 100.0] | 100.0 [83.2 to 100.0] | 100.0 [89.7 to 100.0]
  Week 120: number analyzed (Participants) | 11 | 19 | 30
  Week 120 | 100.0 [71.5 to 100.0] | 100.0 [82.4 to 100.0] | 100.0 [88.4 to 100.0]
  Week 144: number analyzed (Participants) | 6 | 15 | 21
  Week 144 | 100.0 [54.1 to 100.0] | 100.0 [78.2 to 100.0] | 100.0 [83.9 to 100.0]

10. Secondary Outcome: Part 2: Percentage of Male Participants With Maintenance of Suppression of Basal Testosterone to < 30 ng/dL
Description: Male participants with maintenance of suppression of testosterone to < 30 ng/dL are assessed
Time Frame: Weeks 72, 96, 120, and 144
Population: Full analysis set; participants with non-missing observations.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve | Leuprolide Acetate - Overall
Number analyzed (Participants) | 1 | 3 | 4
percentage of participants
  Week 72 | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [39.8 to 100.0]
  Week 96 | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [39.8 to 100.0]
  Week 120 | 100.0 [2.5 to 100.0] | 100.0 [29.2 to 100.0] | 100.0 [39.8 to 100.0]
  Week 144: number analyzed (Participants) | 1 | 1 | 2
  Week 144 | 100.0 [2.5 to 100.0] | 100.0 [2.5 to 100.0] | 100.0 [15.8 to 100.0]

ADVERSE EVENTS:
Time Frame: From screening through end of study; median 949.5 and 1092.0 days for previously-treated and treatment-naïve participants, respectively.
Arm/Group | Leuprolide Acetate - Previously Treated | Leuprolide Acetate - Treament Naïve
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/18 | 1/27
Other Adverse Events (participants affected / at risk) | 18/18 | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Acetate - Previously Treated (N=18) | Leuprolide Acetate - Treament Naïve (N=27)
AFFECTIVE DISORDER (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Leuprolide Acetate - Previously Treated (N=18) | Leuprolide Acetate - Treament Naïve (N=27)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
LYMPHADENOPATHY (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
EAR PAIN (Ear and labyrinth disorders) | 2 (2) | 1 (1)
EYE PAIN (Eye disorders) | 1 (1) | 1 (1)
PHOTOPSIA (Eye disorders) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 3 (4)
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 2 (2) | 0 (0)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 1 (1) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (2) | 3 (3)
HAEMATOCHEZIA (Gastrointestinal disorders) | 1 (1) | 0 (0)
LIP BLISTER (Gastrointestinal disorders) | 1 (2) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 2 (2) | 3 (3)
ORAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTH IMPACTED (Gastrointestinal disorders) | 1 (1) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 2 (2)
VOMITING (Gastrointestinal disorders) | 3 (3) | 3 (5)
CHEST PAIN (General disorders) | 1 (1) | 1 (1)
CRYING (General disorders) | 1 (1) | 4 (4)
FATIGUE (General disorders) | 3 (3) | 0 (0)
FEELING HOT (General disorders) | 2 (2) | 1 (1)
GAIT DISTURBANCE (General disorders) | 1 (1) | 2 (3)
INJECTED LIMB MOBILITY DECREASED (General disorders) | 1 (1) | 0 (0)
INJECTION SITE BRUISING (General disorders) | 2 (2) | 0 (0)
INJECTION SITE DISCOMFORT (General disorders) | 1 (2) | 0 (0)
INJECTION SITE ERYTHEMA (General disorders) | 3 (3) | 4 (4)
INJECTION SITE PAIN (General disorders) | 16 (39) | 26 (94)
INJECTION SITE PRURITUS (General disorders) | 1 (1) | 0 (0)
INJECTION SITE REACTION (General disorders) | 4 (6) | 9 (18)
INJECTION SITE SWELLING (General disorders) | 3 (5) | 1 (2)
INJECTION SITE WARMTH (General disorders) | 3 (3) | 3 (3)
MALAISE (General disorders) | 1 (1) | 0 (0)
MEDICAL DEVICE PAIN (General disorders) | 1 (1) | 0 (0)
PAIN (General disorders) | 5 (9) | 5 (7)
PYREXIA (General disorders) | 6 (6) | 5 (6)
SWELLING (General disorders) | 1 (3) | 2 (2)
TENDERNESS (General disorders) | 2 (2) | 1 (3)
MULTIPLE ALLERGIES (Immune system disorders) | 1 (1) | 2 (2)
SEASONAL ALLERGY (Immune system disorders) | 1 (1) | 2 (2)
COVID-19 (Infections and infestations) | 3 (3) | 9 (10)
GASTROENTERITIS (Infections and infestations) | 3 (3) | 2 (2)
GASTROENTERITIS VIRAL (Infections and infestations) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 4 (5) | 3 (3)
LICE INFESTATION (Infections and infestations) | 1 (1) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 4 (6) | 3 (7)
OTITIS EXTERNA (Infections and infestations) | 1 (1) | 0 (0)
PHARYNGITIS STREPTOCOCCAL (Infections and infestations) | 2 (2) | 4 (6)
SINUSITIS (Infections and infestations) | 1 (1) | 3 (4)
TINEA VERSICOLOUR (Infections and infestations) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 (5) | 7 (8)
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 2 (3)
CONTUSION (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FOOT FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FRACTURED COCCYX (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HAND FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
HUMAN BITE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
NAIL INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
WEIGHT INCREASED (Investigations) | 2 (2) | 0 (0)
ABNORMAL WEIGHT GAIN (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
IRON DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
KNEE DEFORMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 4 (4)
CLUSTER HEADACHE (Nervous system disorders) | 1 (3) | 0 (0)
DIZZINESS (Nervous system disorders) | 0 (0) | 2 (2)
HEADACHE (Nervous system disorders) | 9 (14) | 9 (20)
AFFECTIVE DISORDER (Psychiatric disorders) | 1 (1) | 0 (0)
AGGRESSION (Psychiatric disorders) | 0 (0) | 2 (2)
ANGER (Psychiatric disorders) | 0 (0) | 3 (5)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (1)
ATTENTION DEFICIT HYPERACTIVITY DISORDER (Psychiatric disorders) | 1 (1) | 1 (1)
DEPRESSED MOOD (Psychiatric disorders) | 1 (1) | 0 (0)
EMOTIONAL DISORDER (Psychiatric disorders) | 1 (1) | 5 (7)
HALLUCINATION, AUDITORY (Psychiatric disorders) | 1 (1) | 0 (0)
INITIAL INSOMNIA (Psychiatric disorders) | 0 (0) | 2 (2)
INSOMNIA (Psychiatric disorders) | 2 (2) | 1 (1)
IRRITABILITY (Psychiatric disorders) | 1 (1) | 2 (2)
MOOD ALTERED (Psychiatric disorders) | 1 (3) | 5 (7)
MOOD SWINGS (Psychiatric disorders) | 0 (0) | 2 (2)
TEARFULNESS (Psychiatric disorders) | 1 (1) | 0 (0)
BREAST PAIN (Reproductive system and breast disorders) | 1 (1) | 1 (1)
BREAST TENDERNESS (Reproductive system and breast disorders) | 1 (1) | 1 (2)
NIPPLE PAIN (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
VAGINAL HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 1 (1)
VULVOVAGINAL DISCOMFORT (Reproductive system and breast disorders) | 1 (1) | 0 (0)
VULVOVAGINAL PRURITUS (Reproductive system and breast disorders) | 1 (1) | 1 (1)
BRONCHOSPASM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (5) | 6 (7)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (3)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (3)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 3 (3)
SINUS CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
SNEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
ACNE (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (3)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 3 (3)
SKIN ODOUR ABNORMAL (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
HOT FLUSH (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-08-05): https://cdn.clinicaltrials.gov/large-docs/37/NCT03695237/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT03695237/SAP_001.pdf